CLINICAL TRIAL: NCT06154902
Title: ABE-DESCART Study: Characterization and Outcomes of Patients With Relapsed and Refractory Multiple Myeloma Eligible for Treatment or Treated With Abecma© (Idecabtagene Vicleucel) in Real World Setting in France. A Database Analysis Based on the DESCAR-T Registry
Brief Title: Real-World Outcomes in Relapsed/Refractory Multiple Myeloma Patients Treated, or Eligible for Treatment, With Idecabtagene Vicleucel
Acronym: ABE-DESCART
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA089-1041
Record Dates: First submitted 2023-11-27; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated with idecabtagene vicleucel
  Interventions: Drug: Idecabtagene vicleucel
- Eligible for idecabtagene vicleucel: Eligible for idecabtagene vicleucel treatment but not treated
  Interventions: Other: Not treated

INTERVENTIONS:
Drug: Idecabtagene vicleucel — According to approved product label in France
  Groups: Treated with idecabtagene vicleucel
Other: Not treated — Eligible for idecabtagene vicleucel treatment but not treated
  Groups: Eligible for idecabtagene vicleucel

SUMMARY:
The purpose of this study is to describe demographic and disease characteristics, treatment patterns, and clinical outcomes in the real-world setting among participants in France with relapsed/refractory multiple myeloma (RRMM) who are eligible for treatment with, or have been treated with, idecabtagene vicleucel. This study will use both prospective and retrospective data from the DESCAR-T registry database.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RRMM registered in the DESCAR-T registry and eligible for treatment or treated with idecabtagene vicleucel

Exclusion Criteria:

* Not registered with the social security in France

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in France with RRMM who are eligible for treatment with, or have been treated with, idecabtagene vicleucel
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- DESCAR-T Registry, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html